CLINICAL TRIAL: NCT05049447
Title: Proof of Effectiveness of Pascoflair Using Qantitative Measurement of Electric Brain Activity During Examination Stress in 40 Subjects Suffering From Test Anxiety. A Double-blind, Randomized, Placebo-controlled, 2-armed, Phase IV Study in Parallel Design.
Brief Title: Pharmacological Effects of Pascoflair® on Brain Activity in Patients Suffering From Test Anxiety
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pascoe Pharmazeutische Praeparate GmbH (Industry)
Collaborators: NeuroCode AG (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200S14PF
Record Dates: First submitted 2015-09-21; First posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Stress; Brain Activity; Passiflora Incarnata; Test Anxiety

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum arm (Active Comparator): Intervention: Drug: Verum (Pascoflair)
  Interventions: Drug: Pascoflair
- Placebo arm (Placebo Comparator): Intervention: Drug: Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Pascoflair — 1 x 2 tablets (single-dose)
  Arms: Verum arm
Other: Placebo — 1 x 2 tablets (single-dose)
  Arms: Placebo arm

SUMMARY:
Proof of effectiveness of Pascoflair using qantitative measurement of electric brain activity during examination stress in 40 subjects suffering from test anxiety. A double-blind, randomized, placebo-controlled, 2-armed, Phase IV study in parallel design.

DETAILED DESCRIPTION:
Anxiolytic effects of PASCOFLAIR® shall be tested in subjects suffering from test anxiety after single intake by aid of a newly developed, validated method consisting of a combination of eye tracking (following glances) with neurocode tracking (quantitative EEG with a time resolution of 364 ms).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects.
* Age between 18 and 40 years (both included).
* Anxiety questionnaire PAF (pre-selection of subjects) - values above T> 60 are regarded as conclusive.
* Inconclusive case history and diagnosis.
* Subject must be capable of giving informed consent.
* Acceptance of written consent to participate in the study after education in written and oral form (informed consent).

Exclusion Criteria:

* Acute or chronic disease with an impact on the study, which becomes obvious by case history or clinical examination.
* Clinically relevant pathological findings from clinical and laboratory findings.
* Presence of clinically relevant pathological EEG features or artifact-free portion of the screening EEG <30%.
* Clinically relevant allergic symptoms.
* Detection of alcohol at the time of initial examination (day SC) or on study day A (positive alcohol test) or by case history.
* Detection of drugs (positive drug test) at the time of initial examination (day SC).
* Consumption of clinically relevant medication during last fourteen days before and during the active study period based on the notification of the subject or his case history.
* Consumption of medication with primarily central action (i.e. psychotropic drugs or centrally acting antihypertensives).
* Known intolerance / hypersensitivity (allergy) to plant derived extracts (Passion flower dry extract) or any of the ingredients of the investigational product (anamnestic).
* Presence of a rare, genetic disease such as fructose intolerance, glucosegalactose malabsorption or sucrase-isomaltase deficiency (anamnestic).
* BMI (Body Mass Index) <18 or> 32.
* Consumption of unusual quantities or misuse of coffee (more than 4 cups a day), tea (more than 4 cups a day) or tobacco (more than 20 cigarettes per day).
* Smoking on day of A.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Comparison of verum and placebo Beta 1 power | day A (treatment day) - 1 day
  Comparison of verum and placebo efficacy is performed on electric power in 17 different brain regions within six frequency ranges defined as target parameters in the presence of different stress inducing cognitive tests or exciting video scenes

SECONDARY OUTCOMES:
Tolerability in a 4- Point scale | Final examination (day AB) -1 day
  Tolerability in a 4- Point scale (very good, good, moderately, poor)
Correlation between questionnaire items and spectral EEG power with regard to different frequency ranges. | Final examination - 1 day
  Correlation between questionnaire items and spectral EEG power with regard to different frequency ranges.

IPD SHARING:
Plan to Share IPD: Undecided